CLINICAL TRIAL: NCT02459730
Title: Glass-ionomer Cement Containing Chlorhexidine for ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Aline R F de Castilho, Postdoctoral scholar, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GICCHXART
Record Dates: First submitted 2015-05-13; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Dental Caries
Keywords: Dental caries; glass ionomer cement; ART
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART with GIC containing 1.25% CHX (Experimental): The cavities were filled with the press finger technique using GIC KetacMolar Easymix® containing 1.25% chlorhexidine digluconate (n= 41 tooth surfaces).
  Interventions: Procedure: ART with GIC containing 1.25% CHX.
- ART with GIC (Active Comparator): The cavities were filled with the press finger technique using KetacMolar Easymix® (control group).
  Interventions: Procedure: ART with GIC.

INTERVENTIONS:
Procedure: ART with GIC containing 1.25% CHX. — Carious lesions were prepared by removing infected dentin with hand instruments. No local anesthesia was administered. Then, the cavities were filled with the press finger technique using GIC KetacMolar Easymix® containing 1.25% chlorhexidine digluconate (n= 41 tooth surfaces).
  Arms: ART with GIC containing 1.25% CHX
Procedure: ART with GIC. — Carious lesions were prepared by removing infected dentin with hand instruments. No local anesthesia was administered. Then, the cavities were filled with the press finger technique using KetacMolar Easymix® (n = 66 tooth surfaces).
  Arms: ART with GIC

SUMMARY:
This study evaluated the clinical and microbiological long-term effects of 1.25% CHX associated with GIC applied in primary molars using Atraumatic Restorative Treatment (ART) technique. Randomized controlled trial was conducted on 40 children with carious lesions that received ART either with GIC containing CHX or GIC only. Survival rate of restorations was checked at 3 days, 3 months and 1 year after their placement when the unstimulated saliva samples were collected for microbiological assessment of mutans streptococci (MS) counts. Data were analyzed using ANOVA/Tukey or Kruskal-Wallis/Mann-Whitney tests (p <0.05).

DETAILED DESCRIPTION:
ART treatment and follow-up:

Carious lesions were prepared by removing infected dentin with hand instruments. No local anesthesia was administered. Then, the cavities were filled with the press finger technique with one of the randomly selected materials: (1) GIC KetacMolar Easymix® containing 1.25% chlorhexidine digluconate (KM + CHX; n= 41 tooth surfaces) or (2) KetacMolar Easymix® as a control group (KM; n = 66 tooth surfaces). Material excess was removed using carver instrument and the restoration was coated with a layer of petroleum jelly. Multiple-surface cavities were filled after placement of plastic bands and wedges. Both molars (class I and II) and incisors were treated in this study and the same GIC were used for patients who had more than one carious teeth indicated to ART. The children underwent longitudinal clinical follow-up to assess physical condition (partial or complete fractures) of the restoration and the presence of primary or secondary caries at 7 days, 3 months and 1 year, according to ART evaluation criteria by Frencken et al. Children were encouraged and instructed on dental hygiene and received all other necessary oral care.

Microbiological assays:

Unstimulated whole saliva was collected after 7 days, 3 months and 1 year after treatment from each subject by direct expectoration into a 50-ml sterile container for 5-10 min. Pooled supragingival biofilm samples were collected from all buccal and lingual smooth surfaces, except from the interior of the cavities. In order to standardize plaque amount, a sterile plastic disposable inoculating loop with a circular opening of about 1 µL capacity was used for the collection. Collection was stopped when the opening was filled. Biofilm samples were placed immediately into a 1-ml centrifuge microtubes containing Tris-EDTA buffer (10 mM Tris-Hcl, 0.1 mM EDTA, pH 7.5). Collections were performed at least 1 h after feeding. Tubes were transported on ice to laboratory and processed within 2 h.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* At least one cavitated dentin carious lesion in primary molars or incisors that had an opening wide enough for the smallest ART excavator access

Exclusion Criteria:

* Teeth with pulpal exposure or the presence of fistula and history of pain were excluded

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Clinical long-term effect - Survival Rate | up to 1 year after restorative procedure
  Randomized controlled trial was conducted on 40 children with carious lesions that received ART either with GIC containing CHX or GIC only. Survival rate of restorations was checked after 7 days, 3 months and 1 year of their placement.

SECONDARY OUTCOMES:
Microbiological long-term effect (microbiological assessment of mutans streptococci (MS) counts) | up to 1 year after restorative procedure
  The unstimulated saliva samples were collected for microbiological assessment of mutans streptococci (MS) counts after 7 days, 3 months and 1 year of the dental treatment.